CLINICAL TRIAL: NCT00001415
Title: Glucocorticoid Effects on Cellular Cytokine Release
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940146; 94-M-0146
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-04

CONDITIONS: Depressive Disorder; Fatigue Syndrome, Chronic; Fibromyalgia; Healthy; Inflammation
Keywords: IL-1; IL-6; Immune Response; Inflammation; Steroids; Chronic Fatigue Syndrome; Depression; Fibromyalgia; Normal Volunteer
MeSH Terms: conditions — Depressive Disorder; Fatigue Syndrome, Chronic; Fibromyalgia; Inflammation; Depression

SUMMARY:
A variety of hormones and immune system processes are responsible for how the body responds to illness. This study concentrates on how the hormone cortisol effects the release of immune system factors called cytokines.

Cortisol is a hormone produced in the adrenal glands as a response to stimulation from the pituitary gland. Abnormal levels of cortisol have been seen in several diseases such as depression and multiple sclerosis.

Cytokines are factors produced by certain white blood cells. They act by changing the cells that produce them (autocrine effect), altering other cells close to them (paracrine), and effecting cells throughout the body (endocrine effect). Cytokines are important in controlling inflammation processes.

In this study researchers would like to determine if changes in levels of hormones in the blood are associated with changes in cytokine levels. In addition, researchers would like to learn more about how cytokines respond to hormones in certain diseases.

DETAILED DESCRIPTION:
Many of the biochemical alterations observed in people suffering from major depression are changes in the concentrations and activity of components of the generalized stress response. These include the principal hypothalamic stimulus of pituitary-adrenal activation (corticotropin releasing hormone) and the locus ceruleus/norepinephrine system. The current study attempts to provide a clearer picture of the stability of changes during the acute illness, the treatment phase and the recovery process. We particularly wish to determine whether abnormalities in HPA axis perturbability in the well-state can be demonstrated, and if so how these are related to the acutely-ill state, since this information could provide a quantifiable phenotypic marker for depression.

ELIGIBILITY:
Healthy volunteers.

Depressed patients.

Fibromyalgia patients.

Chronic fatigue patients.

Subjects must not have been treated with steroids for more than two weeks during the previous year.

Subjects must not be on chronic medications.

Subjects must not have known medical problems or any condition which interferes with their immune system's ability to respond to infections (talk with your physician if you are not sure about a particular situation).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130
Dates: Start 1994-05; Study Completion 2000-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] DeRijk RH, Petrides J, Deuster P, Gold PW, Sternberg EM. Changes in corticosteroid sensitivity of peripheral blood lymphocytes after strenuous exercise in humans. J Clin Endocrinol Metab. 1996 Jan;81(1):228-35. doi: 10.1210/jcem.81.1.8550757.
- [Background] Sternberg EM, Chrousos GP, Wilder RL, Gold PW. The stress response and the regulation of inflammatory disease. Ann Intern Med. 1992 Nov 15;117(10):854-66. doi: 10.7326/0003-4819-117-10-854. PMID 1416562